CLINICAL TRIAL: NCT03507270
Title: One-hour Diagnostic Algorithm for Non-ST Elevation Myocardial Infarction Based on Determination of Fatty-acid-binding Protein Concentration
Brief Title: One-hour Diagnostic Algorithm for NSTEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FABP
Record Dates: First submitted 2017-05-22; First posted 2018-04-25 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-05

CONDITIONS: Non ST Segment Elevation Myocardial Infarction
Keywords: FABP; non ST Segment Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Single-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FABP group (Other): Coronary angiography and PCI (according to indications).
  Interventions: Diagnostic Test: FABP

INTERVENTIONS:
Diagnostic Test: FABP — Assessment of changes in FABP concentrations

SUMMARY:
Predictable values of the 1-hour algorithm for estimating the concentration of troponin using highly sensitive reagents are 98-100% for excluding myocardial infarction (MI) and 75-80% for identifying this pathology. Such algorithms are developed for the rapid confirmation or exclusion of myocardial infarction without ST-segment elevation and, when combined with clinical data and electrocardiogram, are used to assess the risk of adverse course of disease and to contribute to decision making about expediency of stay in the intensive therapy unit and early discharge.

In mid-1980s, a new marker of myocardial damage was proposed, namely: fatty-acid-binding protein (FABP). However, the diagnostic value of FABP cannot be interpreted unambiguously because of insufficient number of studies determining the sensitivity and specificity of the test in various manifestations of acute coronary syndrome (ACS).

Available literature presents a wide range of reference values of FABP for MI diagnosis. Reference value ranges are proposed by manufacturers of diagnostic kits based on previous studies. In addition, there is no information about the FABP changes during the first three hours of the disease, as well as there are no data on diagnostic value of changes in this indicator ("∆") in patients with ACS without ST-segment elevation. These considerations provide rationale and support novelty of the planned pilot study.

DETAILED DESCRIPTION:
After enrollment in the study, patients will undergo the following procedures:

1. Physical examination (at baseline) and monitoring of vital signs (blood pressure, heart rate, breathing rate) at hours 1, 2, and 3 after admission to hospital.
2. Registration of 12-lead electrocardiogram (ECG) (at baseline, after 24 hours, and at the day of discharge).
3. At baseline (at the time of admission to hospital), venous blood will be obtained to perform blood tests for determination of troponin I, FABP, and CPK-MB levels. At the same time, venous blood will be sampled for routine clinical laboratory blood tests. At hours 1, 2, and 3 after admission to hospital, venous blood will be sampled for assessment of the troponin I and FABP levels.
4. Echocardiography will be performed 24 hours after admission (LVEDV, LVESV, and EF). At day 3, standard echocardiography will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old
* Male patients
* Acute pain in the chest similar to myocardial infarction with/or without ECG changes
* Admission to the hospital within 4 hours from onset of the disease.

Exclusion Criteria:

* Patients with ACS in the preceding 30 days
* Cerebral blood circulation disorder
* Recent surgical intervention
* Extensive burns of degree 2-3
* Massive wounds and injuries
* Percutaneous coronary intervention or cardioversion
* Pregnancy or lactation
* Malignant tumors of stage 4
* Severe renal insufficiency (GFR< 30 mL/min)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Fatty acid-binding protein (h-FABP) measure | At 4 hours after suspected NSTEMI onset
  Establishing diagnosis of NSTEMI based on h-FABP test for early detection of myocardial infarction

SECONDARY OUTCOMES:
Troponin I (cTnI) measure | At 4 hours after suspected NSTEMI onset
  Establishing diagnosis of NSTEMI based on TnI test
Creatine phosphokinase-MB (CPK-MB) measure | At 4 hours after suspected NSTEMI onset
  Establishing diagnosis of NSTEMI based on CPK-MB test
Creatine phosphokinase (CPK) measure | At 4 hours after suspected NSTEMI onset
  Establishing diagnosis of NSTEMI based on CPK test

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav V. Ryabov, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk NRMC
Locations (1):
- Cardiology Research Institute, Tomsk NRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No